CLINICAL TRIAL: NCT03153566
Title: Comparison Between Tuberculin Vaccine and Cryotherapy in the Treatment of Genital Wart Patients
Brief Title: Comparison Between Tuberculin Vaccine and Cryotherapy in Genital Wart Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mena Ramsis Haleem, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPDG
Record Dates: First submitted 2017-05-12; First posted 2017-05-15 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Genital Wart
MeSH Terms: conditions — Condylomata Acuminata | interventions — Tuberculin; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- study group (Experimental): include (15) patients will be injected with Tuberculin vaccine 0.3 ml every 2 weeks, vaccine will be injected in the largest wart, 4 sessions will be done then patients will be followed for 2 months
  Interventions: Biological: tuberculin
- control group (Active Comparator): include (15) patients will be treated with cryotherapy every 2 weeks ,4 sessions will be done then patients will be followed for 2 months
  Interventions: Device: cryotherapy
- combined group (Experimental): include (15) patients will be treated with combined cryotherapy and Tuberculin vaccine , one week cryotherapy and the other week Tuberculin vaccine , then patients will be followed for 2 weeks
  Interventions: Biological: tuberculin; Device: cryotherapy

INTERVENTIONS:
Biological: tuberculin — inject the mother wart with .3 ml tuberculin vaccine every 2 weeks
  Arms: combined group; study group
Device: cryotherapy — 10 sec 1 cycle into all genital warts
  Arms: combined group; control group

SUMMARY:
Cutaneous and genital warts are common dermatological conditions caused by Human Papilloma Virus. Although it is a benign condition it causes disfigurement, has tendency to collect, can be transmitted to others, this makes adequate and timely treatment important, while many warts are resolve spontaneously over several years, most patients seek treatment because the warts are unsightly and often tender or painful.

DETAILED DESCRIPTION:
Genital warts are highly contagious sexually transmitted diseases (STD) caused by infection of Human Papilloma Virus and, as the most common STD in developed countries, can currently be considered to be globally epidemic.

It is estimated that the frequency of Human Papilloma Virus infection among women in the world ranges from 2% to 44%.

The conventional modalities in treatment of warts include destructive therapies such as salicylic acid, trichloroacetic acid, cryotherapy, silver nitrate, phenol, cantharidin, surgical interventions and laser, antiproliferative agents such as bleomycin, vitamin D analogs, podophyllin, 5 fluorouracil and antiviral agents such as cidofovir and retinoids.

There are different mechanisms have been proposed for the resolution of warts with skin test antigens such as mumps, candida, trichophyton both at the injected as well as distant sites.

Tuberculin:

Purified protein derivative or tuberculin stimulates the cell mediated immunity non specifically by activating T helper 1 cells, Natural Killer cells, and cytokine production an increase in interleukin-12 as a process in boosting the cell-mediated immunity contributes to the mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

* All types of genital and anal warts will be included in this study especially patients with 5 or more warts and more than 1 cm in size

Exclusion Criteria:

* Patients with immunodeficient diseases or receiving any immunosuppressive drugs
* Pregnancy and lactation

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
number of patients with complete resolution of genital warts | 4 months
  frequency (number)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Scott M, Nakagawa M, Moscicki AB. Cell-mediated immune response to human papillomavirus infection. Clin Diagn Lab Immunol. 2001 Mar;8(2):209-20. doi: 10.1128/CDLI.8.2.209-220.2001. No abstract available. PMID 11238198
- [Result] Buck HW Jr. Genital warts. Clin Evid. 2006 Jun;(15):2149-61. No abstract available. PMID 16973081
- [Result] Bosch FX, de Sanjose S. Chapter 1: Human papillomavirus and cervical cancer--burden and assessment of causality. J Natl Cancer Inst Monogr. 2003;(31):3-13. doi: 10.1093/oxfordjournals.jncimonographs.a003479. PMID 12807939
- [Result] Sterling JC, Gibbs S, Haque Hussain SS, Mohd Mustapa MF, Handfield-Jones SE. British Association of Dermatologists' guidelines for the management of cutaneous warts 2014. Br J Dermatol. 2014 Oct;171(4):696-712. doi: 10.1111/bjd.13310. Epub 2014 Oct 1. No abstract available. PMID 25273231
- [Result] Horn TD, Johnson SM, Helm RM, Roberson PK. Intralesional immunotherapy of warts with mumps, Candida, and Trichophyton skin test antigens: a single-blinded, randomized, and controlled trial. Arch Dermatol. 2005 May;141(5):589-94. doi: 10.1001/archderm.141.5.589. PMID 15897380
- [Result] Abd-Elazeim FM, Mohammed GF, Fathy A, Mohamed RW. Evaluation of IL-12 serum level in patients with recalcitrant multiple common warts, treated by intralesional tuberculin antigen. J Dermatolog Treat. 2014 Jun;25(3):264-7. doi: 10.3109/09546634.2013.768760. Epub 2013 May 6. PMID 23336207